CLINICAL TRIAL: NCT06086717
Title: Comparison of Kinesio Taping and Dry Needling in the Management of Grade 1, 2 Knee Osteoarthritis
Brief Title: Comparison of Kinesio Taping and Dry Needling in Grade 1, 2 Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01250 Iram Saeed
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Dry Needling; Joint Flexibility; Kinesio Tape; Knee Osteoarthritis; Pain; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Concurrent Parallel Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Kinesio Taping Group
  Interventions: Other: Kinesio Taping
- Group B (Active Comparator): Dry Needling Group
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Kinesio Taping — One Y-shaped strap with 25% stretch was applied from the mid third of the thigh over the rectus femoris, then its ends directed toward the tibial tuberosity by enwrapping the patella from lateral and medial sides. In 45° knee flexion one eye strap from medial to lateral was applied through the collateral medial and lateral ligaments.
  For the facilitation of VMO 1 eye strap with 25% stretch from medial aspect of thigh to quadriceps tendon. Lastly, 1 eye strap with 25% stretch from tibial tuberosity to lateral aspect of thigh for inhibition of Vastus lateralis
  Arms: Group A
Other: Dry Needling — Following a protocol according to patient and limb, the tensor fasciae latae, hip adductors, hamstrings, quadriceps, gastrocnemius, and popliteus muscles were properly examined in each subject. These muscles are frequently involved in muscle-related knee pain.
  Patients with knee OA who had at least one active MTrP that produced pain were recruited. Patients received a total of 8 DN sessions (2 sessions per week for 4 weeks) at all MTrPs of the lower limbs using the fast-in and fast-out technique (the needle was moved up and down within the muscle).
  Arms: Group B

SUMMARY:
This study's aim was:

- To determine the effects of kinesio taping and dry needling on pain, ROMs, functional mobility, and quality of life in knee OA patients.

DETAILED DESCRIPTION:
This was a randomized clinical trial in which Grade 1, 2 Knee Osteoarthritis patients were randomized into two groups: Group-A and Group-B. Group-A participants received Kinesio taping while Group-B participants received dry needling as an adjunct to the conventional physical therapy treatment. The intervention was carried out for four weeks with frequency of two sessions per week. Outcome measures were assessed at baseline, after two weeks, and after 4 weeks, using Visual Analog Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Knee Range of Motion (ROM), and SF-12 Quality of Life Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed patients of grade 1, 2 knee OA (Kallgren and Lawrence).
* Pain and/or tenderness around knee joint
* Knee OA patients with tightness in Quadriceps, Hamstrings, and Iliotibial band.
* Patients with pain of >4 on VAS.

Exclusion Criteria:

* Patients who had received Intra-articular Steroid injections in knee joints.
* Patients who had suffered a traumatic injury to knee joint within past 6 months prior to this study.
* Patients with any surgical intervention to the knee joints.
* Patients with peripheral vascular disease.
* Patients with diagnosed tumors, malignancies, infection associated with knee joint.
* Patients with lower limb metallic implants.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Pain Score | Baseline, after 2 weeks, and after 4 weeks.
  Pain was measured using Visual Analog Scale on a score from zero (0=no pain) to ten (10=worst pain possible).
Knee ROM | Baseline, after 2 weeks, and after 4 weeks.
  Knee ROM (flexion and extension) was assessed using universal goniometer.

SECONDARY OUTCOMES:
WOMAC Score | Baseline, after 2 weeks, and after 4 weeks.
  Patients' pain, stiffness, and physical functioning of the joints was assessed using WOMAC scale.
Quality of Life Score | Baseline, after 2 weeks, and after 4 weeks.
  Patients health-related quality of life was assessed using SF-12 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University (RIU), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No